CLINICAL TRIAL: NCT00512083
Title: An Open Label Randomized Controlled Dose Escalating Phase II Study of AS1411 Combined With Cytarabine in the Treatment of Patients With Primary Refractory or Relapsed Acute Myeloid Leukemia
Brief Title: Phase II Study of AS1411 Combined With Cytarabine to Treat Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Antisoma Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AS1411-C-201
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Leukemia, Myeloid
Keywords: Leukemia, Myeloid + Acute Disease
MeSH Terms: conditions — Leukemia, Myeloid; Leukemia; Acute Disease | interventions — AGRO 100

INTERVENTIONS:
Drug: AS1411 — AS1411 IV administration continuously over 7 days. Dose either 10mg/kg/day or 40 mg/kg/day.

SUMMARY:
The overall aim of this study is to assess the efficacy and safety of AS1411, over a range of doses, when combined with cytarabine, in the treatment of patients with primary refractory or relapsed acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* primary refractory or relapsed AML
* confirmed diagnosis of AML (de novo or secondary) as defined by WHO classification (Vardiman 2002)
* aged at least 18 years

Exclusion Criteria:

* initial diagnosis of acute promyelocytic leukemia as defined by French-American-British criteria (Bennett 1976)
* patient in blast crisis stage of chronic myeloid leukemia
* received high-dose cytarabine (total cumulative dose of >6g/m sq)in last 6 months
* interval of <6 months between first onset of last complete remission and current relapse
* those with primary refractory leukemia who have received more than three previous induction cycles
* relapsed patients who have received more than three previous treatment regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The prorportion of patients achieving a completel response (CR) after the first cycle of treatment in each treatment group

CONTACTS AND LOCATIONS:
Locations (10):
- United States (9):
  - UCLA Medical Center, Los Angeles, California
  - Univeristy of Colorado Health Cancer Center, Aurora, Colorado
  - St. Francis Hospital and Health Center, Beech Grove, Indiana
  - University of Louisville, James Graham Brown Cancer Center, Louisville, Kentucky
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Duke University Medical Center, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Cancer Therapy and Research Center - Institute for Drug development, San Antonio, Texas
- Christchurch Hospital, Christchurch, New Zealand